CLINICAL TRIAL: NCT00753428
Title: CIDRZ 1236 - Community-based Evaluation of a Pilot PMTCT Project in Kafue District: Impact of HAART to Prevent Pediatric AIDS in Rural Zambia.
Brief Title: Community-based Evaluation of a Pilot PMTCT Project in Kafue District
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0399; X080331005 (Other: UNC)
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Death; HIV Infection
Keywords: HIV-free survival; Community based evaluation; Pregnancy; Under 2 child survival; PMTCT; Pediatric HIV infection; HAART; Routine ART; HIV Seronegativity
MeSH Terms: conditions — Death; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Finger/Heel pricks will be performed for Dried Blood Spot Cards.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Baseline evaluation: Prior to the implementation of the pilot project of giving routine HAART as a method of PMTCT, a minimum of 387 households with children under the age of two will be sampled within each community, for a total of 1,548 households for the first round.
  Interventions: Other: Community-based Survey
- Following implementation: Two years after full implementation of the pilot project of giving routine HAART for PMTCT across all sites, a minimum of 387 households with children under the age of two will be sampled within each community, for a total of 1,548 households. [Note: At time of implementation, we used the same sampling frame for each community. Because of the population increased observed in parts of Kafue, the final number of households significantly exceeded the minimum threshold.]
  Interventions: Other: Community-based Survey

INTERVENTIONS:
Other: Community-based Survey — Questionnaires will be used to record detailed information regarding demographic and socioeconomic characteristics, maternal medical history, recent obstetrical history (including access to preventive services for mother-to-child HIV transmission), and infant medical history. Infant deaths will also be recorded as part of the survey. In cases where either the mother or infant has died, we will perform verbal autopsy interviews (Appendix 5) with surviving family members to determine cause of death and gather information regarding HIV infection and/or exposure.
  Heel/finger pricks will be taken so as to perform dried blood spot cards, and test for HIV in children and adults.

SUMMARY:
In this study, the investigators will assess the population effectiveness of using routine HAART as a PMTCT strategy, through a community-based survey. The survey will be done in the catchment areas of four health clinics in rural Zambia both before and after giving routine ART in the clinics, so as to estimate population HIV-free survival among infants born in each target community.

The investigators hypothesize that incorporation of routine ART into PMTCT will increase the HIV-free survival of exposed infants to 75%.

DETAILED DESCRIPTION:
The primary objective is to determine the incremental benefit of a routine ART strategy for PMTCT on a population basis, when compared to short-course Zidovudine and single-dose Nevirapine (the current PMTCT standard of care).

We will take advantage of planned implementation of a pilot project for routine ART across four primary care centres in rural Zambia (Kafue District). Using a community-based survey modeled after the Demographic and Health Survey, we will measure HIV-free survival among children under two years of age in the catchment areas surrounding these pilot sites, both before and after implementation of services. We will use before-after comparisons in each of these four communities to better understand the incremental benefit of providing these services.

ELIGIBILITY:
Inclusion Criteria:

* Household where a child has been born in the past two years.

Exclusion Criteria:

* Household where there no child has been born in the past two years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Households will be eligible for the full survey if they report that a child was born to a household member within the past two years. If the answer to this question is "yes," an attempt will be made to speak with the mother of the child. If the mother of the child is not available, then the primary care-taker of the child will be interviewed at that time.
Sampling Method: Probability Sample
Enrollment: 4129 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Population HIV-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chi, M.D., Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Reseach in Zambia, Lusaka, Zambia

REFERENCES:
- [Result] Turnbull E, Lembalemba MK, Guffey MB, Bolton-Moore C, Mubiana-Mbewe M, Chintu N, Giganti MJ, Nalubamba-Phiri M, Stringer EM, Stringer JS, Chi BH. Causes of stillbirth, neonatal death and early childhood death in rural Zambia by verbal autopsy assessments. Trop Med Int Health. 2011 Jul;16(7):894-901. doi: 10.1111/j.1365-3156.2011.02776.x. Epub 2011 Apr 7. PMID 21470348
- See also: Website for organisation implementing research study — http://www.cidrz.org/